CLINICAL TRIAL: NCT00466765
Title: Breast Reconstruction and Augmentation With Brava Enhanced Autologous Fat Micro Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brava (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol no. 2004-03
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Mammaplasty; Mastectomy; Lumpectomy
Keywords: Fat Grafting; Breast Augmentation; Liposuctioned Fat Transfer; Lumpectomy; Mastectomy; Micromastia; Asymmetry; Post Lumpectomy Filling Defects; Post implant removal filling defect; Post Mastectomy; Autologous Fat Transfer; Tubular breasts; Tuberous breasts; Constricted breasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Use Brava system for pre-expansion of breast prior to fat grafting
  Interventions: Device: Brava Autologous Fat Transfer System

INTERVENTIONS:
Device: Brava Autologous Fat Transfer System — Number of procedures is based on patient need
  Other Names: Brava System

SUMMARY:
The primary objectives of this study is to determine whether use of a negative pressure external soft-tissue expansion system pre-operatively and post-operatively improves and secures graft survival in autologous fat micro grafting breast augmentation and reconstruction procedures.

DETAILED DESCRIPTION:
Procedure:

Urine pregnancy test will be performed before each designated procedure in the study. Patients will be questioned about underlying renal disease and excluded if existent.

Pre-operative/baseline digital or 35mm photos will be obtained utilizing the standard criteria as performed routinely by plastic and reconstructive surgeons before any surgical procedure. Oblique, frontal and sagittal views will be stored in protected files.

Optional: Patients will have a preoperative breast MRI with the contrasting agent Gadolinium, utilizing a 1.5 Tesla MRI machine and breast coils unless status post breast cancer where no pre-operative MRI is needed. All readings will be performed by board certified radiologists.

Brava domes will be worn bilaterally 3-4 weeks before surgery for 10-12 hours per day, 7 days a week with 24 hour wear for the final 72 hours (3 days) before surgery. Patients will be required to adhere to the dome cleaning process specified by the manufacturer. This is prudent for hygienic reasons and to reduce skin irritation and infections. The domes are for single patient use only. Pressure will range from 15 mmHg to 105mmHg and will be achieved and regulated by either SmartBox, bulb syringe and/or Brava Turbo devices. This will open up the tissue planes and maximally expand the recipient breast in preparation for graft insertion.

Institutional Review Board approval will be obtained and all patients will be properly advised of their rights via signed Informed Consents.

All patients will be assessed by board certified plastic and reconstructive surgeons for autologous fat harvesting sites. Preoperative sedation with IV sedation and/or oral sedation is recommended. Preoperative antibiotics, such as Keflex or similar drug, will be administered before surgery. Sterile drape and prep of the fat harvesting sites will be carried out.

Tumescent anesthetic solution will be prepared by diluting 50cc's of 1% lidocaine with 1/100,000 units of epinephrine with 1000cc's of Ringers Lactate solution and will be instilled with a 14-gauge infusion infiltration cannula into the areas of fat harvesting.

Gentle, low vacuum pressure manual liposuction will be performed to avoid damaging the fat cells. Liposuction will be performed in a standard fashion using 12G & 12 side holes harvesting cannulas and connected to syringes that maintain a controlled constant low vacuum pressure of 300 mmHg (preferably using the K-VAC (Vacuum Assisted Device) syringe). The aspirate will be purged from the syringes into collection bags using atraumatic nonclogging valves (preferably the AT-Valve) or 3 way stopcocks. Once filled, the bags will be spun at low speed (<1000 rpm) to separate fat from serum (and free of oil, if any). The infranatant serum will be drained and the cellular fat supernatant will be concentrated in the bags and directly re-injected into the breasts. Depending upon the volume correction required and the recipient space available, 100 to 500 ml of gently centrifuged (non-packed) fat will be injected per breast.

The recipient breast will be marked carefully prior to infiltration of anesthetics to determine the preferred graft distribution pattern and to select 9-18 graft insertion sites (circumareolar, inframammary, axillary and at the circumference of the breast). The skin will be infiltrated at the graft insertion sites with Naropin 2% (ropivacine).

After the recipient site is anesthetized, puncture sites will be made with a 14-gauge needle. A 14-gauge blunt tip cannula or similar cannula connected to a 3 ml syringe is used to gently inject small droplets distally first and then subsequently proximally as the cannula is withdrawn. Repeated passes at multiple levels in a radial fashion are performed through each of the puncture sites such that the grafts droplets are laid down in a criss-crossing pattern and at multiple planes. Avoid the glandular tissue by remaining in the subcutaneous plane and if more volume is needed and is available proceed to fill the subglandular, intramuscular and submuscular planes. Incision sites are covered with sterile band aids applied to skin. Gentle conforming dressings will be applied to breast.

Elastic garments will be placed on harvest site. Postoperative instructions are handed to each patient. Patient will begin wearing the Brava System, with the SmartBox device only, 18 hours post-operative as a stabilization device. For the first three (3) days the system is worn 24 hours a day or as to the maximum tolerated. If the patient notes pain, the system may be removed and replaced a few hours later. The System is then worn 10 to 12 hours a day for one additional week (7 days). Then the patient may choose to proceed with a prolonged intermittent wear of 10 hours per day for 10 - 14 weeks.

Follow-up will include: A call from the surgical team within 24 hours after surgery. An office follow up visit within 48-72 hours of surgery and follow-up appointment in 6 months. More office follow up visits in the interim are recommended but not mandatory.

A one-year post grafting mammogram will be recommended to all women over the age of 40.

ELIGIBILITY:
Inclusion Criteria:

Female volunteers between the ages of 18 and 80 years of age and weighing between 100- 275 lbs may be enrolled in the study. Ages 16 to 18 with developmental deformities may be enrolled with parental consent.

* Post implant removal with subcutaneous defect
* Post lumpectomy patients with or without radiation therapy with asymmetrical defect
* Post mastectomy with or without radiation therapy
* Post flap reconstruction with asymmetry or contour defect
* Primary breast augmentation
* Primary Post-mastectomy breast reconstruction
* Breast asymmetry
* Other congenital malformation of the breast such as constricted breasts, tubular breast, tuberous breasts, pectus associated deformities and Poland's Syndrome

Exclusion Criteria:

The following volunteers must be excluded from the study:

* A volunteer who has a positive pregnancy test
* A volunteer who has a pacemaker or aneurysm clips
* A volunteer who has had a cardiac stent placed within the last two months
* A volunteer who is claustrophobic
* A volunteer with a known, current substance abuse
* A volunteer with a history of silicone allergy
* A volunteer with a history of Gadolinium allergy (if MRI performed)
* A volunteer with a history of Lidocaine allergy
* A volunteer with a bleeding diathesis
* Untreated breast cancer
* A volunteer who smokes cigarettes or who has a history of smoking within the past three (3) months.
* Medical Conditions including Sever Hypertension, Renal disease, steroid dependant asthma, immuno-suppressed disease, Systemic Lupus, uncontrolled diabetes

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2010-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Digital photographic interpretation by Board Certified Plastic Surgeon or Radiologist. | 6 months

SECONDARY OUTCOMES:
Patient's satisfaction with cosmetic and reconstructive result. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Khouri, MD, Principal Investigator — Brava LLC
Locations (2):
- United States (2):
  - Roger K Khouri, MD, Miami, Florida
  - Miami Breast Center, Medical Office of Roger Khouri MD, Miami, Florida

REFERENCES:
- [Background] Coleman SR, Saboeiro AP. Fat grafting to the breast revisited: safety and efficacy. Plast Reconstr Surg. 2007 Mar;119(3):775-85; discussion 786-7. doi: 10.1097/01.prs.0000252001.59162.c9. PMID 17312477
- [Background] Rigotti G, Marchi A, Galie M, Baroni G, Benati D, Krampera M, Pasini A, Sbarbati A. Clinical treatment of radiotherapy tissue damage by lipoaspirate transplant: a healing process mediated by adipose-derived adult stem cells. Plast Reconstr Surg. 2007 Apr 15;119(5):1409-1422. doi: 10.1097/01.prs.0000256047.47909.71. PMID 17415234
- See also: Information on the Brava System — http://brava.com
- See also: Roger K Khouri, MD information — http://www.miamibreastcenter.com